CLINICAL TRIAL: NCT03068416
Title: CD19-targeting, 3rd Generation CAR T Cells for Refractory B Cells Malignancy - a Phase II Trial.
Brief Title: CD19-targeting, 3rd Generation CAR T Cells for Refractory B Cells Malignancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); AFA Insurance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 004:TCELL; 2016-004043-36 (EudraCT Number)
Record Dates: First submitted 2017-02-21; First posted 2017-03-01 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: B-cell Leukemia; B-Cell Lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR T cells (Experimental): Autologous 3rd generation CD19-targeting CAR T cells
  Interventions: Biological: CAR T cells

INTERVENTIONS:
Biological: CAR T cells — Autologous CD19-targeting, 3rd generation CAR T cells

SUMMARY:
Treatment of patients with B cell lymphoma or leukemia with two doses of CD19-targeting chimeric antigen receptor (CAR) T cells to evaluate for safety and efficacy.

DETAILED DESCRIPTION:
Treatment of patients with B cell lymphoma or leukemia with two doses of CD19-targeting chimeric antigen receptor (CAR) T cells to evaluate for safety and efficacy. The CAR consists of a CD19 targeting antibody scFv with three intracellular signaling domains derived from CD3 zeta, CD28 and 4-1BB. Autologous T cells will be gene engineered with the CAR gene using a retrovirus vector. Prior to T cell infusion, the patients will be subjected to preconditioning treatment. After the second infusion patients will be subjected to immunomodulatory treatment. After T cell infusion, the patients will be evaluated for 24 months for adverse reactions, persistence of CAR T cells and efficacy.

Primary outcome:

- Registration of the safety profile such as inflammation, fever, pain, changes in blood pressure, pulse and other adverse events.

Weekly for the first 6 weeks, then at 3, 6, 9, 12, 15, 18, 21 and 24 months.

Secondary outcome:

Tumor response, CAR T cell persistence and immunological profile

* Determination of tumor size and the tumor marker CD19.
* Determination of the levels of circulating B cells.
* Determination of the level of CAR T cells (mRNA and cells) in blood and biopsies.
* Determination of activation markers on CAR T cells such as CD107a.
* Determination of the presence of immunological markers in blood and biopsies.

At 1 and 3 weeks then at 3, 6, 9, 12, 15, 18, 21 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory CD19+ B-cell lymphoma or leukemia with no other curative treatment option available.
2. Measurable disease.
3. All ages
4. Performance status ECOG 0-2.
5. Fertile females/males must consent to use contraceptives during participation of the trial.
6. Signed informed consent.

Exclusion Criteria:

1. Any significant medical or psychiatric illness that would prevent the patient from giving informed consent or from following the study procedures.
2. Patients with primary CNS lymphoma.
3. Known human immunodeficiency virus (HIV) infection.
4. Active and/or severe infection (e.g. tuberculosis, sepsis and opportunistic infections, active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection.
5. Other serious underlying medical conditions, which, in the Investigator's judgment, could impair the ability of the patient to perform the treatment.
6. Treatment with an investigational product within 30 days prior to enrollment, or at least 5 half-lives of that drug, which is longest.
7. Pregnancy
8. Patients that do not consent to that tissue and blood samples are stored in a biobank
9. Patients whose cells cannot be manufactured.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Safety | 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Tumor response | 24 months.
  Determination of tumor size
B cell levels | 24 months
  Determination of circulating CD19+ B cells
CAR T cell persistence | 24 months
  Determination of the level of CAR T cells
Immunological profile | 24 months
  Determination of frequencies of immune cells in patient blood and tissues
Cytokine profile | 24 months
  Determination of cytokine profile in patient blood

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Enblad, MD, PhD, Principal Investigator — Uppsala University Hospital, Dept of Oncology
Locations (1):
- Uppsala University Hospital, Dept of Oncology, Uppsala, Sweden

REFERENCES:
- [Derived] Saren T, Ramachandran M, Gammelgard G, Lovgren T, Mirabello C, Bjorklund AK, Wikstrom K, Hashemi J, Freyhult E, Ahlstrom H, Amini RM, Hagberg H, Loskog A, Enblad G, Essand M. Single-Cell RNA Analysis Reveals Cell-Intrinsic Functions of CAR T Cells Correlating with Response in a Phase II Study of Lymphoma Patients. Clin Cancer Res. 2023 Oct 13;29(20):4139-4152. doi: 10.1158/1078-0432.CCR-23-0178. PMID 37540566